CLINICAL TRIAL: NCT05472337
Title: Effect of Colchicine on Coronary Reperfusion in Patients With Acute Coronary Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210507002
Record Dates: First submitted 2022-05-23; First posted 2022-07-25 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Colchicine; Myocardial Infarction; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Acute Coronary Syndrome; Myocardial Reperfusion; Anti-Inflammatory Agents
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Infarction; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Prospective randomized comparison between colchicine versus no colchicine in terms of microvascular coronary reperfusion and infarct size in patients with acute coronary syndrome.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Colchicine (Experimental): Subjects allocated to the intervention group will receive colchicine + standard of care for 6 weeks.
  Interventions: Drug: Colchicine
- Standard of Care - Control (No Intervention): Subjects allocated to the control group will receive only standard of care for 6 weeks.

INTERVENTIONS:
Drug: Colchicine — Oral colchicine (1 mg loading dose followed by 0.5 mg 1 hour later, administered 6 to 24 hours before angioplasty, followed by 0.5 mg (1 comp.) per day for 6 weeks.
  Arms: Colchicine

SUMMARY:
This randomized clinical trial will determine the treatment effect of colchicine (1.5 mg loading dose and 0.5 mg daily thereafter) for 6 weeks on microvascular coronary reperfusion and infarct size in patients with acute coronary syndrome.

DETAILED DESCRIPTION:
Despite significant advances in the treatment of coronary artery disease, acute coronary syndromes (ACS) remain one of the leading causes of mortality and morbidity worldwide. In Chile, it is estimated that cardiovascular disease is responsible for one out of every four deaths Moreover, the consequences of an infarction, i.e., myocardial damage and death, lead to disability, loss of productivity, and economic costs.

Based on the knowledge that ACS occurs as a consequence of the atheroma plaque complication (rupture or erosion) and the consequent thrombosis at that level, current therapy in patients admitted for ACS includes :

(i) acute inhibition of thrombosis by means of antiplatelet and anticoagulant drugs.

ii) Coronary revascularization for severe stenosis by means of coronary angioplasty or bypass surgery.

These therapies have resulted in marked patient benefit, however, in many cases fail to reduce myocardial damage and to achieve adequate myocardial reperfusion.

In fact, in up to 50% of patients with ACS undergoing angioplasty inadequate myocardial reperfusion is observed, despite achieving correct repermeabilization of the coronary artery.

The complication of an atheromatous plaque leading to ACS results from the presence of inflammatory cells, which weaken the vessel wall and promote thrombosis. Both monocytes and neutrophils are key in these phenomena. By intervening in the plaques by means of angioplasty - which includes balloon and implantation of high-pressure stents - both plaque debris, thrombi, and inflammatory cells are released into microcirculation.

This triggers an inflammatory response at this level, which promotes endothelial and tissue edema, myocardial hemorrhage, and direct occlusion of these microvessels.

The result is that even with an adequate recanalization of the epicardial coronary artery (which has the complicated plaque) tissue reperfusion is insufficient, complicating proper recovery of the affected myocardium.

Colchicine is a low-cost, safe, widely available, anti-inflammatory drug, with multiple uses in cardiovascular pathology.

It is recommended in patients with acute pericarditis, including those post-infarction, and has recently been shown to be useful in preventing new cardiovascular events in patients with ACS. Previous studies have shown that during coronary angioplasty in patients with ACS, inflammatory cytokines, neutrophil-derived microparticles, and Neutrophil Extracellular Traps (NETS) are released into the microcirculation.

These are recognized as key agents in the No-Reflow phenomena, by promoting inflammation facilitating thrombosis, and occluding microvessels. Our studies have also shown that the use of Colchicine in a single dose 6 to 24 hours prior to coronary angioplasty results in a dramatic reduction in the release of these inflammatory cytokines and NETs at the time of coronary angioplasty.

It is possible then, that Colchicine is potentially a new strategy to prevent No-Reflow associated with coronary angioplasty in patients with ACS.

In addition, a recent sub-analysis of the Colchicine Cardiovascular Outcomes Trial (COLCOT study, which assessed the use of colchicine vs. placebo in patients with ACS) showed that the use of colchicine mainly benefited those patients who initiated it within the first 3 days of their event and resulted in significantly fewer cardiovascular (CV) episodes (cardiovascular death, infarction, stroke, or emergency hospitalization for angina) at 2-year follow-up, compared with those who initiated it later.

IMR has been shown to have prognostic implications in ACS patients undergoing angioplasty.

The higher the value, the higher the microvascular obstruction, resulting in less myocardial recovery. Index of Microvascular Resistance (IMR) can, in fact, independently predict left ventricular function and infarct size and it is considered a therapeutic target and a relevant measurement in determining the prognosis of patients. Therefore, measurement of IMR before and after angioplasty, makes it possible to determine changes in microcirculation related to the procedure.

Therefore, investigators aim to conduct an open-label randomized controlled trial to evaluate the effects of adding colchicine to standard care among patients with acute coronary syndrome in terms of microvascular obstruction after coronary angioplasty in patients with ACS, as measured by the IMR.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Adults hospitalized at the Clinical Hospital of the Catholic University for an ACS condition, defined as:

   - Presence of chest pain, associated with enzymatic elevation (increase of ultrasensitive troponin above normal value (99th percentile)) with or without electrocardiographic changes.
3. Patients undergoing coronary angiography with the intention of angioplasty in the next few days (during the index hospitalization).
4. Ability and willingness to provide written informed consent.

Exclusion Criteria:

1. ST-segment elevation myocardial infarction (undergoing emergency angioplasty therefore not allowing time for the administration and effect of colchicine).
2. Severe left main stenosis.
3. Advanced heart failure, left ventricular ejection fraction <35%.
4. Related to colchicine use: known intolerance, previous use for another condition (e.g., gout), severe liver disease (e.g., severe liver disease).
5. Severe liver disease (transaminase elevation 3 times above normal), blood dyscrasia (leukocyte or platelet count lower than normal), glomerular filtration rate (MDRD), use of CYP3A4 or calcineurin inhibitors, active autoimmune disease or the use of chronic anti-inflammatory therapy, concomitant infection, pregnancy or concomitant infection, pregnancy or lactation.
6. Any other disease that limits life expectancy to <1 year.
7. Medical history of a disorder that could, in the opinion of the treating physician, place the participant at significant risk if they were to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in Index of Microcirculatory resistance (IMR) between pre and post-coronary angioplasty. | baseline ( pre-angioplasty) and at the end of the procedure (angioplasty)
  Invasive assessment of Index of Microvascular Resistance (IMR) before and after angioplasty in both colchicine and control group.

SECONDARY OUTCOMES:
Average value of endpoint IMR. | at the end of the procedure (angioplasty)
  Comparison of IMR obtained post- angioplasty between colchicine and control group
Change in cardiac enzyme levels (troponin) before and after angioplasty in both colchicine and control group. | baseline (pre-angioplasty) and 24 h post-angioplasty
  Measurement of Troponin before and after angioplasty in both colchicine and control group
Change in level of inflammatory markers ( Ultra-sensible C-reactive protein and IL-6) at baseline and 6 week follow-up. | baseline (prior to Colchicine administration) and at 6 weeks after discharge
  Measurement of Ultra-sensible C-reactive protein and Interleukin-6 before and after angioplasty in both colchicine and control group
Percent of salvaged myocardium. | baseline (two - four days post-angioplasty and at 6 weeks after discharge
  Measurement of salvaged myocardium using cardiac magnetic resonance imaging in both colchicine and control group

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Martínez, MD, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Hospital Clínico Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No